CLINICAL TRIAL: NCT01421615
Title: Effect of Different Courses of Lactobacilli Treatment on Bacterial Vaginosis and Related Pregnancy Outcomes
Brief Title: Effect of Different Courses of Lactobacilli Treatment on Bacterial Vaginosis and Pregnancy Outcomes
Acronym: BV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Li Yanfang, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GZ board of health
Record Dates: First submitted 2011-08-08; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial vaginosis; Probiotics; Lactobacilli; Pregnancy outcome; Randomized controlled trial
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lotion (Placebo Comparator): lotion:the patients in control group receive washing medicine and are followed up to the 4rd～7th days of postpartum.
  Interventions: Drug: Vaginal capsules of lactobacilli
- lactobacilli capsule (Experimental)
  Interventions: Drug: Vaginal capsules of lactobacilli
- lactobacilli capsules (Experimental)
  Interventions: Drug: Vaginal capsules of lactobacilli

INTERVENTIONS:
Drug: Vaginal capsules of lactobacilli — The patients in one-course group who were BV positive would receive the first course treatment of vaginal lactobacillus capsule and be repeatedly evaluated BV status after treatment. If their BV test result were still positive after one-course treatment, they would NOT receive any treatment but would be followed up to the 4th-7th days of postpartum.
  Other Names: Brand names: Dingjunsheng; Commodity code name: A246912309879; Approved by the state: S20030005
Drug: Vaginal capsules of lactobacilli — The patients in two-course group who were BV positive would receive the first course treatment of vaginal lactobacillus capsule and be repeatedly evaluated BV status after treatment. If their BV test result were still positive after one-course treatment, they will receive the second course treatment of Lactobacilli preparation.
  Other Names: Brand names: Dingjunsheng; Commodity code name: A246912309879; Approved by the state: S20030005
  Arms: lactobacilli capsule; lotion

SUMMARY:
The purpose of this study is to examine the effect of lactobacillus preparation on Bacterial vaginosis (BV) in low-risk pregnant women and to evaluate the value of double courses for the patients with durative positive result. It is assumed that the living preparation of lactobacillus was beneficial for treatment of BV during pregnancy. The two-courses treatment can increase the response rate and improve pregnancy outcomes in the durative BV positive patients comparing with one-course one.

DETAILED DESCRIPTION:
Research method: This was a single-blind randomized controlled trial.

Diagnostic standard: The study population is the women who have positive outcome of screened test for BV by sialidase method.

Allocation and follow up: Patients who were screened for BV by sialidase method and randomly allocated into control group、one-course group and two-course group. The patients in control group who were BV positive would receive lotion washout and be repeatedly evaluated BV status per two weeks and be followed up to the 4th～7th days of postpartum. The patients in one-course group and in two-course group who were BV positive would receive the first course treatment of vaginal lactobacillus capsule and be repeatedly evaluated BV status after treatment. The patients in two-course group will receive the second course treatment of Lactobacilli preparation if their BV test result were still positive after one-course treatment, but those in one-course group would NOT receive any treatment even though they would have the durative BV positive result after one-course of Lactobacilli. The patients in the two interventional groups would be repeatedly evaluated BV status at 28th gestational weeks and be followed up to the 4th-7th days of postpartum. All the inspection results of vaginal secretions and pregnancy outcome were recorded.

Outcome measures:

* The prevalence of BV,the response rates of lactobacillus preparation,the recurrence rate.
* The adverse pregnancy outcomes of mother.
* The adverse pregnancy outcomes of perinatal fetus.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at 16-18 gestational weeks with no history of premature labor or premature rupture of fetal membranes.

Exclusion Criteria:

* who have menstrual disorder or forget the last menstrual period, and have no type-B ultrasonic result, so the gestational week is not clear.
* Who have monilial vaginitis, trichomonas vaginitis, or sexual transmitted diseases.
* who have severe medicochirurgic diseases.
* multiple pregnancy.
* anomalies of genital tract
* fetal anomaly

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5000 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who transformed to negative status of bacterial vaginosis | 6 months
  The patients who were BV positive would receive treatment and be repeatedly evaluated BV status on the time of post-treatment 1 week, 28th gestational weeks, and before birth, respectively.The number of Participants who transformed to negative status of bacterial vaginosis will be recorded. The rates of bacterial vaginosis transformed to negative status will be calculated.

SECONDARY OUTCOMES:
pregnancy outcome of mother | 6 months (from 16~18 gestational weeks to the 4th-7th days of postpartum)
  1. the delivery weeks
  2. the delivery mode
  3. the presence of premature rupture of fetal membra
  4. the presence of premature labor
  5. the volume of postpartum haemorrhage
  6. the presence of pregnancy complications
  7. the highest temperature during the first three days of postpartum
pregnancy outcome of perinatal fetus | 6 months (from 16~18 gestational weeks to the 4th-7th days of postpartum)
  1. the neonatal birth weight
  2. the presence of fetal distress
  3. the neonatal 1 min Apgar score
  4. the numerically highest value of neonatal transcutaneous bilirubinometry
Safety and tolerability | 6 months (from 16~18 gestational weeks to the 4th-7th days of postpartum)
  1. liver function test
  2. renal function test

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Lee, Master, Principal Investigator — The First Affiliated Hospital of Guangzhou University of TCM
Locations (1):
- Maternal and child care hospital in Panyu District, Guangzhou, Guangdong, China